CLINICAL TRIAL: NCT02643251
Title: A Multicenter, Randomized, Double Blind, Parallel-Group Study Comparing the Efficacy and Safety of Clonidine Hydrochloride Topical Gel, 0.1%, to Clonidine Hydrochloride Gel Comparator in the Management of Painful Diabetic Neuropathy
Brief Title: The Efficacy and Safety of Clonidine Hydrochloride Topical Gel, vs Clonidine Hydrochloride Gel Comparator to Treat Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLO-291
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Painful Diabetic Neuropathy; Diabetic Neuropathy; Neuropathy
Keywords: Diabetes Mellitus; Pain; Foot Pain; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine Hydrochloride Topical Gel,0.1% (Experimental): Clonidine Hydrochloride Topical Gel,0.1%
  Interventions: Drug: Clonidine Hydrochloride Topical Gel, 0.1%
- Clonidine Hydrochloride Gel Comparator (Placebo Comparator): Clonidine Hydrochloride Gel Comparator
  Interventions: Drug: Clonidine Hydrochloride Gel Comparator

INTERVENTIONS:
Drug: Clonidine Hydrochloride Topical Gel, 0.1% — Clonidine Gel is supplied as an aqueous gel formulation for topical use.
  Other Names: Clonidine Gel
  Arms: Clonidine Hydrochloride Topical Gel,0.1%
Drug: Clonidine Hydrochloride Gel Comparator — Clonidine Gel Comparator is supplied as an aqueous gel formulation for topical use.
  Other Names: Clonidine Gel Comparator
  Arms: Clonidine Hydrochloride Gel Comparator

SUMMARY:
The study will include three (3) phases: Screening Phase, Treatment Phase, and Follow-up Phase. Subjects who qualify to participate will apply study drug to their feet three times daily and will record their daily pain scores using an interactive voice response system (IVRS) during the Treatment Phase for 12 weeks. Approximately 100 adult subjects will be randomized to receive Clonidine Gel or Clonidine Gel Comparator.

DETAILED DESCRIPTION:
Study CLO-291 is a randomized, double-blind, comparator-controlled, parallel-group, multicenter study of 0.1% clonidine topical gel (Clonidine Gel) for the treatment of pain associated with painful diabetic neuropathy. The study will include three (3) phases: Screening Phase, Treatment Phase, and Follow-up Phase. Subjects who satisfy all eligibility criteria will apply Clonidine Gel Comparator to their feet three times daily and will record their daily pain scores using an interactive voice response system (IVRS). Approximately 100 adult subjects will be randomized to receive Clonidine Gel or Clonidine Gel Comparator during the 12 week Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is fluent in English and has provided written informed consent.
2. Subject is an outpatient ≥18 years of age at the time of the Screening Visit.
3. Subject has Type 1 or Type 2 diabetes mellitus with a hemoglobin A1C value < 10% and has been stable on therapy (diet, oral anti-hyperglycemic, and/or insulin) for at least six (6) months prior to the Screening Visit.
4. Subject is a male or non-pregnant, non-lactating female. Females must be practicing an acceptable method of birth control or be surgically sterile or postmenopausal (amenorrhea for ≥12 months). A negative pregnancy test at the Screening and Day 1 visits is required for females of child-bearing potential. Double-barrier methods, hormonal contraceptives, and abstinence are acceptable birth control methods for this study.
5. Subject has chronic pain attributable to a symmetrical stocking distribution neuropathy in the lower extremities for at least six (6) months. Pain should be clearly localized to the area of neuropathy (feet), and subjects should be able to distinguish the target pain from other painful areas and conditions.
6. Subject has an average pain score relevant to the target pain in the feet of ≥4 on an 11 point numerical pain rating scale over the previous 24 hours at the Screening Visit.
7. Subject meets a pre-specified, minimum numerical pain rating scale score following capsaicin skin challenge.
8. Subject must satisfactorily complete Accurate Pain Reporting and Minimizing Placebo Response Training.
9. Subject must have moderate to severe pain during the Screening Run-in Phase.
10. Subjects must be 75 to 110% compliant with application of study drug during the Screening Run-in Phase
11. Subject has been medically stable for at least 30 days prior to the Screening Visit, and in the opinion of the Investigator, is in otherwise good general health based on medical history, physical examination, electrocardiogram, and laboratory evaluation.

Exclusion Criteria:

1. Subject has neuropathy secondary to non-diabetic causes in the opinion of the Investigator (e.g., vasculitis, familial neuropathy, alcoholism, pernicious anemia, hepatitis, malignancy, chronic inflammatory demyelinating polyneuropathy [CIDP], human immunodeficiency virus [HIV], medication-induced neuropathy, vitamin B12 deficiency).
2. Subject has a significant neurological disorder or condition that might confound assessment of painful diabetic neuropathy (e.g., stroke with distal neurological deficit, mononeuritis multiplex, lumbar radiculopathy).
3. Subject has a confounding disorder as determined by the Algorithm for Excluding Disorders that Masquerade as Painful Diabetic Neuropathy.
4. Subject has other sustained pain with intensity at or greater than the bilateral neuropathic pain in the feet.
5. Subject is using an implanted medical device (e.g., spinal cord stimulator, intrathecal pump, or peripheral nerve stimulator) for treatment of pain.
6. Subject is hypotensive with a resting diastolic blood pressure <60 mm Hg or a systolic blood pressure <90 mm Hg at the Screening or Day 1 Visit.
7. The subject has recent history (within the past 3 months) or current symptoms of orthostatic hypotension.
8. Subject has a history of foot or toe amputation or an active foot or toe ulcer.
9. Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study.
10. Subject has a history of substance abuse disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, within the past year, has current evidence of substance abuse disorder, is receiving medical treatment for drug abuse, or has a positive urine drug screen for a non-prescribed substance of abuse.
11. Subject is receiving or has received within 30 days prior to the Screening Visit any prohibited medications or is anticipated to receive after the start of the trial any new prescription medication for their painful diabetic neuropathy. Subjects may be enrolled if stable on therapy for painful diabetic neuropathy.
12. Subject has symptomatic or severe coronary insufficiency, clinically significant cardiac conduction disturbances, myocardial infarction (within last 12 months), moderate to severe cerebrovascular disease, or severe chronic obstructive pulmonary disease (COPD).
13. Subject has estimated creatinine clearance less than 50 mL/min (Cockcroft Gault) at the Screening Visit.
14. Subject has serum alanine transaminase (ALT) or aspartate transaminase (AST) >3.0 times the upper limit of normal or total bilirubin concentrations >2.0 times the upper limit of normal at the Screening Visit.
15. Subject has received an investigational drug within 30 days prior to the Screening Visit.
16. Subject has been treated previously with clonidine topical gel or participated in a clonidine topical gel clinical study, including Study CLO 290.
17. Subject is currently taking or has taken clonidine (any formulation) over the past 4 weeks.
18. Subject has known hypersensitivity or intolerance to clonidine.
19. Subject is receiving or has received ≤7 days prior to the start of the Screening Phase "alternative medicine" products or treatments (e.g., acupuncture, naturopathy, homeopathy, etc.) for management of pain.
20. Subject has a history of malignancy within the past 5 years except for successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix.
21. Subject is planning to have surgery during the course of the study.
22. Subject has significant skin changes on physical examination associated with either pedal edema or venous stasis disease.
23. Subject has any dermatologic condition of the lower extremities that could affect study drug absorption
24. Subject has current symptoms of depression with a Beck Depression Inventory II (BDI II) score >19 at the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Shaibani, MD, Principal Investigator — Nerve and Muscule Center of Texas
Locations (23):
- United States (23):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Norco, California
  - Sacramento, California
  - Santa Monica, California
  - Tustin, California
  - Fort Myers, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Blackfoot, Idaho
  - Boise, Idaho
  - Belleville, Illinois
  - Blue Island, Illinois
  - Chicago, Illinois
  - Hazelwood, Missouri
  - Cleveland, Ohio
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Clonidine Hydrochloride Topical Gel, 0.1%: Clonidine Hydrochloride Topical Gel, 0.1%
  Clonidine Hydrochloride Topical Gel, 0.1%: Clonidine Gel is supplied as an aqueous gel formulation for topical use.
Period: Overall Study
Arm/Group | Clonidine Hydrochloride Topical Gel, 0.1% | Clonidine Hydrochloride Gel Comparator
Started | 69 | 69
Completed | 58 | 67
Not Completed | 11 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — PI Decision to terminate patient | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine Hydrochloride Topical Gel, 0.1% | Clonidine Hydrochloride Gel Comparator | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 47 | 98
  >=65 years | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.76) | 59.7 (10.00) | 59.5 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 54 | 54 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 24 | 42
  White | 49 | 43 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 84 (Week 12) in Numeric Pain Rating Scale Score
Description: The Numeric Pain Rating Scale is a single reading that measures the patients interpretation of their pain on a scale from 0, no pain to 10, worst pain imaginable. The change from baseline can range from -10 to 10. The change from Baseline (averaged over Day -14 to Day -8) to End-of-Treatment (averaged over Days 78 to 84 [±3 days]) in the Numeric Pain Rating Scale score assessing the "average pain in the past 24 hours in the painful areas of the feet" averaged over Days 78 to 84 compared to the 7 days at the Baseline Phase (Days -14 to -8). For the primary efficacy endpoint, the mean change in pain intensity from Baseline to Week 12 was analyzed using an analysis of covariance (ANCOVA) model with the Baseline pain intensity score serving as a covariate. The statistical model also included treatment, site, site by treatment interaction, and strata. If the site by treatment interaction term was not significant at the 0.1 level, then it was excluded from the model.
Time Frame: The change from Baseline (averaged over Day -14 to Day -8) to End-of-Treatment (averaged over Days 78 to 84 [±3 days])
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clonidine Hydrochloride Topical Gel, 0.1% | Clonidine Hydrochloride Gel Comparator
Number analyzed (Participants) | 58 | 68
units on a scale | -1.2 (1.395) | -1.4 (1.526)
Statistical Analysis 1: Comparison: Clonidine Hydrochloride Topical Gel, 0.1% vs Clonidine Hydrochloride Gel Comparator; Test type: Superiority; p = 0.3361, Mixed Models Analysis

2. Secondary Outcome: Mean Daily Worst Pain Intensity Numeric Pain Rating Scale Scores
Description: The Numeric Pain Rating Scale is a single reading that measures the patients interpretation of their pain on a scale from 0, no pain to 10, worst pain imaginable. The change from baseline can range from -10 to 10. The change from Baseline (worse score from Day -14 to Day -8) to End-of-Treatment (worse score during Days 78 to 84 [±3 days]) in the Numeric Pain Rating Scale score assessing the "worse pain in the past 24 hours in the painful areas of the feet" from Days 78 to 84 compared to the 7 days at the Baseline Phase (Days -14 to -8). For the primary efficacy endpoint, the mean change in pain intensity from Baseline to Week 12 was analyzed using an analysis of covariance (ANCOVA) model with the Baseline pain intensity score serving as a covariate. The statistical model also included treatment, site, site by treatment interaction, and strata. If the site by treatment interaction term was not significant at the 0.1 level, then it was excluded from the model.
Time Frame: The change from Baseline (worse over Day -14 to Day -8) to End-of-Treatment (worse over Days 78 to 84 [±3 days])
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clonidine Hydrochloride Topical Gel, 0.1% | Clonidine Hydrochloride Gel Comparator
Number analyzed (Participants) | 58 | 68
units on a scale | -1.29 (1.734) | -1.48 (1.667)

ADVERSE EVENTS:
Arm/Group | Clonidine Hydrochloride Topical Gel, 0.1% | Clonidine Hydrochloride Gel Comparator
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/69 | 6/69
Other Adverse Events (participants affected / at risk) | 4/69 | 2/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Hydrochloride Topical Gel, 0.1% (N=69) | Clonidine Hydrochloride Gel Comparator (N=69)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Perirectal absess (Infections and infestations) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Hydrochloride Topical Gel, 0.1% (N=69) | Clonidine Hydrochloride Gel Comparator (N=69)
Headache (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days